CLINICAL TRIAL: NCT02388828
Title: Long-term Follow-up of Subjects Exposed to Lentiviral-based CART-meso Gene Therapy Products in Cancer Studies
Brief Title: CART-meso Long-term Follow-up
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 33514, 821715; 821715 (Other: UPenn)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Subjects Who Have Received Lentiviral-based CART-meso Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects who have received lentiviral-based CARTmeso therapy
  Interventions: Biological: lentiviral-based CART meso therapy

INTERVENTIONS:
Biological: lentiviral-based CART meso therapy

SUMMARY:
This is a non-therapeutic, long-term follow-up (LTFU) study of subjects who have received retroviral-based gene therapy products in cancer studies. All subjects in this LTFU protocol have received lentiviral modified T cells engineered to express an anti-mesothelin scFv Chimeric Antigen Receptor (CAR). This gene therapy product is called CART-meso. Lentiviruses are a subfamily of retroviruses. This protocol is designed in adherence with the November 2006 Food and Drug Administration (FDA) Guidance for Industry, "Monitoring for Delayed Adverse Events" and "Supplemental Guidance on Testing for Replication Competent Retrovirus in Retroviral Vector Based Gene Therapy Products and During Follow-up of Patients in Clinical Trials Using Retroviral Vectors " and involves up to 15 years of monitoring of subjects who have been exposed to retrovirus-mediated gene transfer. Subjects will undergo biannual visits for a blood test evaluating persistence of cells with retroviral vector sequences, chemistry, hematology and tumor markers (as applicable). On annual visits, subjects will further undergo a physical exam and medical history (including concomitant medications and adverse events) with careful attention to features possibly related to retrovirus-induced diseases

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be enrolled into this destination protocol because they have received CART-meso cells that were genetically modified with a lentiviral vector. All subjects who have participated in a lentiviral vector study under IND #15882 and have received CART-meso cells will be asked to participate in this protocol.
* Subjects 18 years of age and older
* Subjects who have provided informed consent prior to their study participation.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have received lentiviral-based CARTmeso therapy
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | At each visit until study completion, up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Haas, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No